CLINICAL TRIAL: NCT03067246
Title: A Comparison of Two Supraglottic Devices, the VBM Intubating Laryngeal Tube and I-Gel
Brief Title: A Comparison of the VBM Intubating Laryngeal Tube and the I-Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16LO1210
Record Dates: First submitted 2016-12-16; First posted 2017-03-01 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2018-02

CONDITIONS: Airway Management
Keywords: Supraglottic device; Fibre optic scope; Endotracheal intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VBM Intubating Laryngeal Tube (Active Comparator): Device: VBM Intubating Laryngeal Tube Intervention: VBM Intubating Laryngeal Tube insertion, seal pressure, endotracheal intubation
  Interventions: Device: VBM Intubating Laryngeal Tube
- I-Gel (Active Comparator): Device: I-Gel Intervention: I-Gel insertion, seal pressure, endotracheal intubation
  Interventions: Device: I-Gel

INTERVENTIONS:
Device: VBM Intubating Laryngeal Tube — The position of the VBM Intubating Laryngeal Tube will be assessed using a fibreoptic scope following balloon inflation of the cuff. Seal pressure will be assessed with the presence of the inflated cuff. Endotracheal intubation through the intubating laryngeal tube with a size 7 VBM reinforced tube will be assessed using a fiberoptic scope.
  Arms: VBM Intubating Laryngeal Tube
Device: I-Gel — The position of the I-Gel will be assessed using a fibreoptic scope. The seal pressure will be assessed with the specified design of the I-Gel in the absence of a cuff. Endotracheal intubation through the I-Gel with a size 7 reinforced endotracheal tube will be assessed using a fiberoptic scope.
  Arms: I-Gel

SUMMARY:
A study comparing two second generation supraglottic Airway devices, the VBM intubating laryngeal tube and the I-Gel.

DETAILED DESCRIPTION:
This is a study comparing the use of a newer generation laryngeal mask to the 2nd generation widely used at present. The company responsible for the manufacture of this product is VBM Medizintechnik GmBH, Germany. The recent difficult airway society guidelines recommend the use of these newer generation devices and this has been the incentive to conduct this project. These newer generation supraglottic devices have an additional feature which is an extension of the mask with a balloon that sits in the oesophagus. The trial is investigating ease of placement of these devices, ventilatory pressures, leak pressure and ease of intubation through the VBM device compared to I-Gel. The position of the supraglottic device on insertion and the position of the endotracheal tube will be confirmed with a fibrescope. A follow up will take place on the same day and after 24 hours for symptoms of a sore throat postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient between the age of 18 - 70
2. Any patient having the capacity to consent
3. Any patient requiring general anaesthesia but not endotracheal intubation immediately after induction of anaesthesia.

Exclusion Criteria:

1. Patient refusal
2. Patients involved in another research project
3. Patients who require endotracheal intubation immediately after induction of anaesthesia
4. Patients who are systemically unwell/unstable
5. Patients at risk of aspiration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Time in seconds required for placement of supraglottic device | Through study completion, an average of 30 minutes
  Time from device first enters mouth and appearance of end-tidal CO2

SECONDARY OUTCOMES:
Seal pressure measured in cmH2O | Through study completion, an average of 30 minutes
  Peak seal pressure when manual ventilation is commenced
Successful endotracheal intubation through the supraglottic airway, end tidal carbon dioxide monitoring in kilopascals | Through study completion, an average of 30minutes
  This is performed with the endotracheal tube mounted onto the fibreoptic scope and placed through the supraglottic device. The patients will be extubated immediately following the end of the surgical procedure which may take an average of approximately 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Ahmad, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available

REFERENCES:
- [Result] Miller DM. Third generation supraglottic airways: is a new classification needed? Br J Anaesth. 2015 Oct;115(4):634-5. doi: 10.1093/bja/aev310. No abstract available. PMID 26385673
- See also: Link to correspondence relating to the article — https://doi.org/10.1093/bja/aev310